CLINICAL TRIAL: NCT06404905
Title: A First-in-Human, Open Label, Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Antitumor Activity of BT02 in Patients With Advanced Solid Tumors
Brief Title: Clinical Trial of BT02 in Patients With Advanced Solid Tumors
Acronym: BT02
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT02-101
Record Dates: First submitted 2024-03-19; First posted 2024-05-08 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumors

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BT02 treatment (Experimental): BT02 given intravenously administer in patients with advanced solid tumors.
  Interventions: Drug: BT02 monoclonal antibody injection

INTERVENTIONS:
Drug: BT02 monoclonal antibody injection — It is expected to include 10-30 patients assigned to dose escalation cohorts.

SUMMARY:
A First-in-Human, Open Label, Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Antitumor Activity of BT02 in Patients with Advanced Solid Tumors

DETAILED DESCRIPTION:
Overall study design:

This is an open-label, FIH, Phase I / II study of BT02 to evaluate the safety, tolerability, PK, immunogenicity, and preliminary antitumor activity of BT02 in adult patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 at the time of signing the informed consent form, male or female;
2. Patients must have histologically or cytologically confirmed diagnosis of advanced solid tumor;
3. Adequate organ and hematologic function;
4. Patients must have at least measurable or evaluable lesion in phase I and measurable lesion in phase II according to RECIST 1.1;
5. ECOG performance status 0~1;
6. Life expectancy ≥ 3 months;
7. Good compliance and be willing to follow-up visit.

Exclusion Criteria:

1. Receive treatment before study as below:

   a) Previous systematic anti-cancer therapy;
2. Active or prior documented autoimmune disease within past 2 years;
3. History of clinically significant cardiovascular disease;
4. Significant acute or chronic infections;
5. Prior toxicities from anti-cancer therapies have not regressed to grade ≤1 severity;
6. Any prior Grade≥3 irAE while receiving immunotherapy;
7. Unstable brain metastasis or meningeal metastasis with clinical symptoms;
8. Patients with mental disorders or poor compliance;
9. Known alcohol or drug abuse;
10. Other severe systemic diseases or conditions that unsuitable for participating in this study in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | Within day 28 after administration
  safety
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | Within day 28 after administration
  Safety
Maximum tolerated dose | Within day 28 after administration
  Maximum tolerated dose

SECONDARY OUTCOMES:
The Pharmacokinetics characteristics of BT02 | Within day 28 after administration
  Levels of BT02 in blood
Progression-free survival (PFS) | From date of enrollment until the date of revocation of informed consent, termination from the trial, or initiation of new anti-tumor treatment, loss of follow-up or death, whichever came first, assessed up to 100 months.
  The time from the date of first study treatment to the first occurrence of disease progression.
Overall survival (OS) | From date of enrollment until the date of revocation of informed consent, termination from the trial, or initiation of new anti-tumor treatment, loss of follow-up or death, whichever came first, assessed up to 100 months.
  The time from the date of first study treatment to death from any cause.
Duration of response | From date of enrollment until the date of revocation of informed consent, termination from the trial, or initiation of new anti-tumor treatment, loss of follow-up or death, whichever came first, assessed up to 100 months.
  The time from first occurrence of a documented response to disease progression.
Objective Response Rate (ORR) | From date of enrollment until the date of revocation of informed consent, termination from the trial, or initiation of new anti-tumor treatment, loss of follow-up or death, whichever came first, assessed up to 100 months.
  The sum of the proportion of subjects with CR or PR

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Beijing, Biejing, China

IPD SHARING:
Plan to Share IPD: No